CLINICAL TRIAL: NCT00585767
Title: Functional, Dynamic, and Anatomic MR Urography
Status: Withdrawn | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200311391
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hydronephrosis
Keywords: Hydronephrosis
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with two kidneys
- 2: Patients with solitary kidney

SUMMARY:
This is a clinical feasibility study to assess the value of MR imaging for obtaining functional, dynamic and anatomical information in a comprehensive imaging protocol in subjects having obstructive uropathy.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older.
* All female patients of childbearing potential must agree to use a medically accepted method of contraception at the time of the study.
* Patients must have the ability to understand the requirements of the study, provide written and informed consent to participate, and agree to abide by the study requirements.
* Patients who have known or suspected hydronephrosis or patients with solitary kidneys.

Exclusion Criteria:

* Patients with known or suspected hypersensitivity to gadolinium-based agents.
* Patients who are pregnant or lactating.
* Patients with a condition that is a contraindication to MRI (e.g., cardiac pacemaker, epicardial pacemaker leads, cochlear implants, ferromagnetic aneurysm clip, ferromagnetic halo device, or other conditions that would preclude patient proximity to a strong external magnetic field).
* Patients with a recent history of hemolytic anemia, sickle cell anemia or other hemoglobinopathy.
* Patients with a history of significant claustrophobia.
* Patients with impaired renal function based on 24-hr urine collection (creatinine clearance <10 ml/min or serum creatinine >1.8 mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with obstructive uropathy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2001-04; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Katzburg, MD, Principal Investigator — University of California, Davis